CLINICAL TRIAL: NCT00355186
Title: SWiss Multicenter Intracoronary Stem Cells Study in Acute Myocardial Infarction (SWISS-AMI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Roberto Corti, MD, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWISS-AMI
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Acute Myocardial Infarction
Keywords: acute myocardial infarction; MRI; bone marrow cells; stem cells; remodeling

ARMS (3):
- Control (No Intervention)
- Early (Experimental)
  Interventions: Procedure: intracoronary bone marrow cells infusion
- Late (Experimental)
  Interventions: Procedure: intracoronary bone marrow cells infusion

INTERVENTIONS:
Procedure: intracoronary bone marrow cells infusion — intracoronary bone marrow cell infusion via a OTW balloon; "Stop-flow-technique" as previously described
  Arms: Early; Late

SUMMARY:
Title: SWiss multicenter Intracoronary Stem cells Study in Acute Myocardial Infarction (SWISS-AMI).

Study population: Patients with acute myocardial infarction, treated with primary PCI.

Objective: To determine whether intracoronary infusion of BMCs improves recovery of left ventricular function after acute myocardial infarction treated by PCI

Design: Multi-center, randomized, controlled clinical trial with central core lab analysis for MRI.

Therapy: Intracoronary infusion of BMCs in the infarct related artery at 5-7 days or 3-4 weeks after successful primary PCI

Primary Endpoint: Change in global left ventricular ejection fraction (LVEF) at 4 months relative to baseline measured by quantitative MRI.

Secondary Endpoints:

* Change in LVEF at MRI at 12 months
* Change in regional left ventricular wall motion and thickness at 4 and 12 months.
* Change in infarct size at 4 and 12 months as assessed by "delayed enhancement" technique by MRI
* Analysis of the myocardial infarct size and transmurality, time to PCI and coronary flow characteristics after PCI as predictor of LV remodeling and change after cell therapy
* Change in myocardial perfusion at 4 and 12 months
* Change in serum level of amino-terminal pro-brain natriuretic peptide (NT pro-BNP)
* Major adverse cardiac events (MACE: death, myocardial infarction, TVR (ACBP or PCI, stroke, hospitalization for cardiac reasons) at 12 months

Interventions:

* Aspiration of 50 ml bone marrow (<24 hours) prior to administration
* Intracoronary balloon-based infusion of 10 ml BMCs
* Cardiac MRI at baseline (resp. at hospital discharge), at 4 and 12 months

Therapy groups: Bone marrow-derived stem cells infusion in the successfully revascularized infarct related vessel at day 5-7 or day 21-28.

Control group: Management according to the "state of the art" medical therapy after successful primary PCI.

Safety: A study independent "safety committee" will analyze the clinical results after the first 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* Visual LVEF at angiogram or echocardiography ≤45%
* Treatment by primary PCI within 24 hours of the onset of chest pain or initial treatment with thrombolysis within the 12 hours followed by PCI within the 24 hours of the onset of chest pain
* Significant regional LV wall motion dysfunction in the infarct related territory
* Age >18 years

Exclusion Criteria:

* Abnormal regional wall motion outside the infarct region
* Known previous myocardial infarction in the same target vessel
* Known pre-existing left ventricular dysfunction (EF<45% prior to admission)
* Need for revascularization in the non infarct-related coronary within 4 months
* Pre-existing symptoms of heart failure or known cardiomyopathy
* Known active infection or chronic infection with HIV, HBV or HCV
* Chronic inflammatory disease
* Serious concomitant disease with a life expectancy of less than one year
* Follow up impossible (no fixed abode, etc)
* Contraindication for cardiac MRI (i.e. pace maker, neurostimulator, claustrophobia)
* Severe renal failure (creatinine >250 mmol/l)
* Relevant liver disease (GOT > 2x norm or spontaneous INR > 1,5)
* Anemia (Hb < 8.5 mg/dl), Thrombocytopenia (<100.000/µl)
* Pregnancy
* Participation at a clinical trial in the last 30 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-08; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in global left ventricular ejection fraction (LVEF) at 4 months relative to baseline measured by quantitative MRI | 4 months

SECONDARY OUTCOMES:
Change in LVEF at MRI at 12 months | 12 months
Change in regional left ventricular wall motion and thickness at 4 and 12 months | 4 and 12 months
Change in infarct size at 4 and 12 months as assessed by "delayed enhancement" technique by MRI | 4 and 12 months
Analysis of the myocardial infarct size and transmurality transmurality, time to PCI and coronary flow characteristics after PCI as predictor of LV remodeling and change after cell therapy | baseline 4 and 12 months
Change in myocardial perfusion at 4 and 12 months | 4 and 12 months
Change in serum level of amino-terminal pro-brain natriuretic peptide (NT pro-BNP) | 4 and 12 months
Major adverse cardiac events (MACE: death, myocardial infarction, TVR (ACBP or PCI, stroke, hospitalization for cardiac reasons) at 12 months | 4 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Corti, MD, Principal Investigator — Cardiology, University Hospital Zurich, Switzerland; Thomas F Luescher, MD, Study Chair — Cardiology, University Hospital Zurich
Locations (4):
- Switzerland (4):
  - Cardiology, University Hospital Berne, Bern
  - Kantonsspital, Lucerne
  - Cardiocentro Ticino, Lugano
  - Cardiology, university Hospital Zurich, Zurich

REFERENCES:
- [Derived] Gastl M, Surder D, Corti R, Faruque Osmany DMM, Gotschy A, von Spizcak J, Sokolska J, Metzen D, Alkadhi H, Ruschitzka F, Kozerke S, Manka R. Effect of intracoronary bone marrow-derived mononuclear cell injection early and late after myocardial infarction on CMR-derived myocardial strain. Int J Cardiol. 2020 Jul 1;310:108-115. doi: 10.1016/j.ijcard.2020.01.025. Epub 2020 Jan 15. PMID 31982162
- [Derived] Surder D, Manka R, Moccetti T, Lo Cicero V, Emmert MY, Klersy C, Soncin S, Turchetto L, Radrizzani M, Zuber M, Windecker S, Moschovitis A, Buhler I, Kozerke S, Erne P, Luscher TF, Corti R. Effect of Bone Marrow-Derived Mononuclear Cell Treatment, Early or Late After Acute Myocardial Infarction: Twelve Months CMR and Long-Term Clinical Results. Circ Res. 2016 Jul 22;119(3):481-90. doi: 10.1161/CIRCRESAHA.116.308639. Epub 2016 Jun 6. PMID 27267068
- [Derived] Surder D, Gisler V, Corti R, Moccetti T, Klersy C, Zuber M, Windecker S, Moschovitis A, Kozerke S, Luscher TF, Erne P, Manka R. Thrombus formation in the left ventricle after large myocardial infarction - assessment with cardiac magnetic resonance imaging. Swiss Med Wkly. 2015 Jun 22;145:w14122. doi: 10.4414/smw.2015.14122. eCollection 2015. PMID 26098589
- [Derived] Surder D, Manka R, Lo Cicero V, Moccetti T, Rufibach K, Soncin S, Turchetto L, Radrizzani M, Astori G, Schwitter J, Erne P, Zuber M, Auf der Maur C, Jamshidi P, Gaemperli O, Windecker S, Moschovitis A, Wahl A, Buhler I, Wyss C, Kozerke S, Landmesser U, Luscher TF, Corti R. Intracoronary injection of bone marrow-derived mononuclear cells early or late after acute myocardial infarction: effects on global left ventricular function. Circulation. 2013 May 14;127(19):1968-79. doi: 10.1161/CIRCULATIONAHA.112.001035. Epub 2013 Apr 17. PMID 23596006
- [Derived] Surder D, Schwitter J, Moccetti T, Astori G, Rufibach K, Plein S, Lo Cicero V, Soncin S, Windecker S, Moschovitis A, Wahl A, Erne P, Jamshidi P, Auf der Maur C, Manka R, Soldati G, Buhler I, Wyss C, Landmesser U, Luscher TF, Corti R. Cell-based therapy for myocardial repair in patients with acute myocardial infarction: rationale and study design of the SWiss multicenter Intracoronary Stem cells Study in Acute Myocardial Infarction (SWISS-AMI). Am Heart J. 2010 Jul;160(1):58-64. doi: 10.1016/j.ahj.2010.03.039. PMID 20598973